CLINICAL TRIAL: NCT04985240
Title: Randomized Intervention Study With Crop Lettuce Enriched With Molybdenum
Brief Title: Intervention Study on Molibdenum Biofortification Vegetables ( Nutri-Mo-Food )
Acronym: NutMoFood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Sonya Vasto, Associate professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Nutri-Mo-Food2021
Record Dates: First submitted 2021-07-18; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Healthy Diet
Keywords: functional food; molibdenum

STUDY DESIGN:
Intervention Model Description: The study were designed by two cohorts The control group and the interventional group. The intervention lasted for 10 days and 100gr of lettuce per day was consumed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: (control group) (Experimental): The control group was assigned to crop lettuce without any biofortification but with the same characteristic of bioforticated lettuce(soil, water, harvesting time).
  Interventions: Dietary Supplement: Lettuce with no biofortification
- Experimental: intervention group (Experimental): The intervention group was assigned to biofortificated Molibdenum crop lettuce.
  Interventions: Dietary Supplement: Intervention Molibdenum group

INTERVENTIONS:
Dietary Supplement: Lettuce with no biofortification — Lettuce without any biofortification was assigned to each participant belonging to the control group which ate 100gr every day for 10 days
  Arms: No Intervention: (control group)
Dietary Supplement: Intervention Molibdenum group — Lettuce with Iodine biofortification was assigned to each participant belonging to the intervention group which ate 100gr every day for 10 days
  Arms: Experimental: intervention group

SUMMARY:
The aim of the project is to study of the influence of Lettuce crop enriched with Molibdenum on hematological parameter. Secondary outcome to find out Molibdenum presence in urine in order to evaluate vegetables, like little crop, as Molibdenum biocarrier.

DETAILED DESCRIPTION:
everal human pathologies are caused by deficiencies of some mineral elements. These deficiencies can be overcome through careful dietary diversification and mineral supplementation. An alternative or even complementary way is represented by the intake of bio-fortified foods. In the field of mineral deficiency increasing the bioavailable mineral concentration in vegetables intended for human consumption; can be a useful tool to prevent many harmful pathologies. Therefore, in this scenario, it appears very important to identify the right dosages and the most effective methods of administration to bio-fortify vegetables with a strong nutritional-health connotation.

The present project aim to investigate the benefits of fortified food intake in a cohort of healthy individuals. Specifically, we have fed healthy individuals with lettuce enriched with Molibdenum and collected plasma and urine samples after 7-10 days. Each subject was subjected to two venous blood samples taken at the beginning of the observation and at the end. The samples thus obtained will be transported in certified containers for the safe transport of biological samples, and, subsequently, processed by the experimenters at the laboratories of the Molecular Biology section of the University of Palermo. Serum and plasma will be obtained from each blood sample. All information thus obtained will be recorded in a database in which each person will be identified with a numerical code, in order to comply with current privacy regulations. Body weight, Barefoot standing height, Body mass index, Body composition will be measured in the different groups of study. Samples will be analyzed and compared for glucose, albumin, total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides, uric acid, creatinine, AST, ALT, γ-GT, ALP, bilirubin, Ferritin, free Iron, transferrin, total proteins, Magnesium, Calcium, insulin, osteocalcin, hematocrit, hs-CRP, Bone metabolism (Osteocalcin, parathyroid hormone, CTX, Calcitonin), Vitamin D Calcium, Phosphate, Potassium, gastric hormones ( GIP, GLP1, GLP2, ghrelin, glucagon, PYY, CCK) oxidative stress markers (LDL-ox, AGE, urinary 8-iso-prostaglandin F (PGF)2alpha) and inflammatory markers(IL-1, TNF, IL-6, IL-10)

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* age: 18-65 years
* healthy status
* no drug therapy or integration therapy

Exclusion Criteria:

* Inflammatory chronic disease
* use of medication or suffering from any condition
* pregnancy
* breastfeeding
* current smokers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Urine Molibdenum concentration (mg/l) | 10 days
  Urine Molibdenum concentration (mg/l) will be assessed at baseline and after 10 days
Haematology and serum chemistry measurements | 10 days
  glucose, albumin, total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides, uric acid, creatinine, AST, ALT, γ-GT, ALP, bilirubin, Ferritin, free Iron, transferrin, total proteins, Magnesium, Calcium, insulin, Vitamin D Calcium, HCRP, Potassium, Phosphate, will be assessed at baseline and after 10 days

SECONDARY OUTCOMES:
Body mass Index (BMI) kg/m2 | 10 days
  Weight (Kg), height (M), BMI (kg/m2) All these measurements will be assessed at baseline and after 10 days
body composition | 10 days
  lean mass as percent of body weight and fat mass as percent of body weight will be assessed at baseline and after 10 days
Gastric Hormones (pg/ml) | 10 days
  GIP(pg/ml), GLP1(pg/ml), GLP2(pg/ml), ghrelin(pg/ml), glucagon(pg/ml), PYY(pg/ml), CCK(pg/ml) measured in plasma will be assessed at baseline and after 10 days
Oxidative stress marker (ng/mL) | 10 days
  LDL-ox (ng/mL), AGE (ng/mL), urinary 8-iso-prostaglandin F (PGF)2alpha (ng/mL) measured in plasma will be assessed at baseline and after 10 days
Inflammatory markers (ng/ml) | 10 days
  IL-1 (ng/ml), TNF(ng/ml), IL-6(ng/ml), IL-10(ng/ml) measured in plasma will be assessed at baseline and after 10 days
Bone metabolism markers (pg/mL) | 10 days
  Osteocalcin(pg/mL), parathyroid hormone(pg/mL), CTX, Calcitonin(pg/mL) measured in plasma will be assessed at baseline and after 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biological, Chemical and Pharmaceutical Sciences and Technologies, Palermo University, Palermo, PA, Italy